CLINICAL TRIAL: NCT03651141
Title: The Effects of Myofascial Decompression and Neurodynamic Sliding on the Hamstring for Division I Track and Field Athletes With Hamstring Tightness
Brief Title: The Effects of Soft Tissue Therapy and Exercise on Hamstring Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Principal Investigator, Samantha Wagner, Principal Investigator, Graduate Student, Oklahoma State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ED174
Record Dates: First submitted 2018-03-29; First posted 2018-08-29 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hamstring Tightness; Myofascial Pain; Musculoskeletal Pain
Keywords: Hamstring tightness; myofascial decompression; cupping; neurodynamic sliding
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neurodynamic Sliding (Experimental): neurodynamic sliding consists of 2 movements; 1) movement 1 involves sitting on the edge of the treatment table the bringing their neck to their chest along with bending their knee and pointing their ankle to the ground. Movement 2 is performed by facing their head towards the ceiling and straightening their knee while pointing their ankle towards their nose. Subjects will alternate these 2 active movements for 60s and repeated 5 times, with rest period of 15s between sets.
  Interventions: Other: Neurodynamic Sliding
- Myofascial Decompression (Experimental): For the group receiving the cupping treatment, the subject will lay on their stomach and their affected hamstring will be exposed. Cocoa butter will be applied to the hamstring prior to the application of the cups. 5 cups will be placed along the hamstring and calf muscles. Using a handheld suction pump, each cup will be pumped so that skin fills up half of the cup. The cups will stay in place for five minutes and the clinician will instruct the subject to perform 5 repetitions of active quad sets and 5 repetitions of ankle pumps .
  Interventions: Other: Myofascial Decompression
- Diathermy (Sham Comparator): The control group will receive a sham heat (diathermy treatment). The subjects will be asked to sit and relax for five minutes and the machine will not be turned on with a timer timing the treatment.
  Interventions: Other: Diathermy

INTERVENTIONS:
Other: Neurodynamic Sliding — Subjects in the neurodynamic sliding group perform 2 movements; 1) movement 1 involves sitting on the edge of the treatment table the bringing their neck to their chest along with bending their knee and pointing their ankle to the ground. Movement 2 is performed by facing their head towards the ceiling and straightening their knee while pointing their ankle towards their nose. Subjects will alternate these 2 active movements for 60s and repeated 5 times, with rest period of 15s between sets. A metronome will be set at 30 beats per minute for 15 full slides per minute to standardize the amount of slides per session.
  Arms: Neurodynamic Sliding
Other: Myofascial Decompression — For the group receiving the cupping treatment, the subject will lay on their stomach and their affected hamstring will be exposed. Cocoa butter will be applied to the hamstring prior to the application of the cups. 5 cups will be placed along the hamstring and calf muscles. Using a handheld suction pump, each cup will be pumped so that skin fills up half of the cup. The cups will stay in place for five minutes and the clinician will instruct the subject to perform 5 repetitions of active quad sets and 5 repetitions of ankle pumps .
  Arms: Myofascial Decompression
Other: Diathermy — The control group will receive a sham heat (diathermy treatment). The subjects will be asked to sit and relax for five minutes and the machine will not be turned on with a timer timing the treatment.
  Arms: Diathermy

SUMMARY:
The purpose of this study is to investigate the effects of myofascial decompression (cupping) and neurodynamic sliding technique for the hamstring on Division I Track and Field athletes who complain of hamstring tightness. Research questions will be: how do these techniques affect hamstring range of motion and flexibility; isometric strength of the hamstring muscle; muscle activation; and rate of force development. The hypotheses of this study are that neurodynamic sliding will have an effect on all variables and myofascial decompression will only have an effect on range of motion.

DETAILED DESCRIPTION:
Predisposing factors to hamstring injury include neural tension and muscle flexibility restrictions due to fascial adhesions. The sciatic nerve can produce symptoms of pain, decreased range of motion, and increased resting muscle tone when it is overstretched. The nerve can be overstretched after a hamstring injury and cause adhesions on the nerve and abnormal mechanosensitivity leading to perceived hamstring tightness.The purpose of this study is to investigate the effects of myofascial decompression (cupping) and neurodynamic sliding technique for the hamstring on Division I Track and Field athletes who complain of hamstring tightness. Research questions will be: how do these techniques affect hamstring range of motion and flexibility; isometric strength of the hamstring muscle; muscle activation; and rate of force development. The hypotheses of this study are that neurodynamic sliding will have an effect on all variables and myofascial decompression will only have an effect on range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Must be in the Sprints, Jumps, or Multi (heptathlon, pentathlon, or decathlon) groups
* complain of hamstring tightness and/or injury in the last calendar year
* have less than 80⁰ for Active Knee Extension test.

Exclusion Criteria:

* Past history or current neurological disorders or orthopedic diseases
* Surgery of the lower extremity that involves an autograft on the tested leg
* Past history of hamstring surgery
* Receiving current treatment for a hamstring injury
* Received any form of myofascial therapy or neurodynamic techniques within the last week unhealed wounds
* active TB
* leukemia
* hemophilia
* thrombocytopenia
* fever
* influenza
* moderate/severe anemia
* high blood pressure
* cardiac conditions
* late stages of pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
Hamstring Flexibility change | Baseline, 5 minutes after intervention, and within 24 hours of intervention
  Using the 'Active Knee Extension test', subjects are placed supine with both the hip and knee positioned at 90° of flexion and then asked to extend lower leg until point of limitation. A digital inclinometer is used to measure the angle of the knee joint in this position to examine flexibility of the hamstring muscle group.

SECONDARY OUTCOMES:
Hamstring muscle strength change | Baseline, 5 minutes after intervention, and within 24 hours of intervention
  Peak torque production of the hamstring muscles will be assessed using an isokinetic dynamometer with the subjects performing a maximum voluntary isometric contraction with the knee in a slightly flexed position.
Time of Force Development | Baseline, 5 minutes after intervention, and within 24 hours of intervention
  Time to reach peak force torque
Electromyographic (EMG) Muscle Activation of the Hamstring muscles | Baseline, 5 minutes after intervention, and within 24 hours of intervention
  The electrical activation signaling of the hamstring muscles will be measured using electromyography during the isometric contraction.
Disablement of the Physically Active patient outcome survey | Baseline, 5 minutes after intervention, and within 24 hours of intervention
  The Disablement of the Physically Active Scale (DPAS) paper survey will be used to assess subject perceptions of impairment, limitation, disability and quality of life related to their hamstring discomfort. The scale ranges from 0 (No disability) to 64 (Severe disability) in which the scores will be compared.
Functional Patient Outcome survey | Baseline, 5 minutes after intervention, and within 24 hours of intervention
  The Lower Extremity Functional Scale is a questionnaire containing 20 questions about a subject's ability to perform everyday tasks. Scores range from 0-4 and represent 'extreme difficulty' or 'unable to perform activity' to 'no difficulty'. The maximum score on the survey is 80 points, with lower total scores indicating a greater perceived disability.

CONTACTS AND LOCATIONS:
Overall Officials: Aric Warren, EdD, Study Chair — Oklahoma State University
Locations (1):
- Applied Neuromuscular Physiology Lab, Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No